CLINICAL TRIAL: NCT00393588
Title: The Use of Magnetic Resonance Imaging to Investigate Cortical Damage in Patients With Multiple Sclerosis and Correlation With Cognitive Dysfunction
Brief Title: Magnetic Resonance Imaging to Detect Brain Damage in Patients With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070014; 07-N-0014
Record Dates: First submitted 2006-10-27; First posted 2006-10-30 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-09-29

CONDITIONS: Multiple Sclerosis
Keywords: Brain; Cognitive Deficits; Cognitive Testing; MRI; Multiple Sclerosis; MS; Healthy Volunteer; HV
MeSH Terms: conditions — Multiple Sclerosis; Cognition Disorders

SUMMARY:
This study will test the ability of magnetic resonance imaging (MRI) to detect damage in different parts of the brain in patients with multiple sclerosis and to see if cognitive problems in patients can be correlated with the presence of lesions or reduction in the size of certain part of the brain. Healthy subjects will also be studied to compare findings in patients with those of normal volunteers.

Healthy subjects and patients with multiple sclerosis who are between 18 and 60 years of age may be eligible for this study. Patients must not have severe clinical disability and must have been receiving and responding to Interferon beta for at least 6 months prior to enrollment. Candidates are screened with a medical history, physical examination, MRI and possibly evoked potential testing, which measures the nervous system response to visual, auditory and somatosensory stimulation.

Participants have two MRI scans within 1 week (inclusive of the one performed for screening). MRI uses a magnetic field and radio waves to obtain images of body tissues and organs. The scanner is a metal cylinder surrounded by a strong magnetic field. During the MRI, the subject lies on a table that can slide in and out of the cylinder. Participants will be tested with magnet strengths of 1.5 and 3 Tesla; the higher the Tesla, the greater the ability to see brain changes. Each scan may last up to 90 minutes. In addition to the MRI scans, participants undergo cognitive testing that measures memory and thought processes and complete forms that test and quantify fatigue level, stress, anxiety and depression

DETAILED DESCRIPTION:
OBJECTIVE: The study will evaluate cognitive impairment in patients with multiple sclerosis (MS) and correlate the degree of cognitive dysfunction as identified by scores obtained in multiple cognitive tests with measurements of cortical thickness, cortical lesions and white matter disease on magnetic resonance imaging of brains of MS individuals.

STUDY POPULATION: Study population will consist of 49 patients with relapsing remitting or secondary progressive MS with superimposed relapses who have been treated with Interferon beta at fully tolerated dosages for at least six months, and 49 healthy volunteers matched for gender, age and educational level. We expect to screen 65 individuals per arm in order to be able to enroll 49 individuals per arm, thus meeting the requirements of the sample size calculations.

DESIGN: After screening clinical (rating disability by the means of the Expanded Disability Status Scale [EDSS] score), neurophysiological (e.g. evoked potential tests) and imaging examinations, MS patients and healthy subjects will undergo a neuropsychological evaluation using the Minimal Assessment of Cognitive Function in Multiple Sclerosis (MACFIMS) and the Automated Neuropsychological Assessment Metrics (ANAM), and also a 3 Tesla magnetic resonance imaging (MRI). After 25% and after 50% of projected patients have been enrolled, distribution in MACFIMS will be evaluated to ensure that a broad spectrum of cognitive ability is represented. Cortical thickness, cortical lesions and white matter damage metrics (e.g. lesion load, diffusion tensor and magnetization transfer MRI measures) will be computed. In order to exclude the hypothesis that the presence of fatigue, anxiety and depression, normally occurring in MS patients, might interfere with their cognitive performance, thus acting as confounding factors, scales measuring fatigue and mental status will be administered in all subjects. Scores obtained on these scales will be used as covariates in each of the statistical analyses performed in the present study to account for their possible effects.

OUTCOME MEASURES: The first outcome measure will be the MACFIMS and cortical thickness values. Correlation between these two metrics will be initially performed. Secondly, cortical lesions as well as white matter lesions on T1 and T2 weighted images, magnetization transfer ratios and diffusion tensor imaging metrics of lesional and normal appearing brain tissues will be computed and their impact in determining cognitive impairment will be determined. Thirdly, deep gray matter, white matter and total brain volume measures will be computed and correlated with cognitive function measured by the MACFIMS. Similarly, correlations between clinical disability, as measured by the EDSS score and cognitive impairment, as well as between EDSS score and each of the RMI variables explored in the study will be performed. Finally, the level of correlation between MACFIMS and ANAM tests will be investigated.

ELIGIBILITY:
* PATIENT INCLUSION CRITERIA:
* Diagnosis of relapsing remitting or secondary progressive with superimposed relapses MS.
* Age between 18 and 60, inclusive.
* EDSS between 0 and 6.5.
* Receiving treatment with Interferon beta (either 1a or 1b) at fully tolerated dose for at least 6 months prior to enrollment and with evidence of clinical efficacy (i.e. reduction or absence of clinical relapses) at the time of the enrollment.

PATIENT EXCLUSION CRITERIA:

* Clinical relapse at the time of the enrollment or within the previous 3 months.
* Undergoing chronic therapy with any other immunomodulatory or immunosuppressive medication (excluding standard dosages of steroids intravenously/intramuscularly injected and orally taken for the treatment of relapses) besides Interferon within the past 6 months.
* Currently taking medications used for treatment of cognition/fatigue such as Donepezil (Aricept), Modafinil (Provigil), Amantadine, or other drugs that may act as temporary stimulants or depressants for the central nervous system.
* Currently taking other medications used for symptomatic relief that may affect cognition. The study neurologist will make the determination of eligibility.
* Clinically significant medical condition that, in the opinion of the investigator, would compromise patient's safety or affect his/her MRI (e.g., diabetes mellitus, chronic hypertension, severe anemia, kidney disease, heart disease [angina, arrhythmias, congestive heart failure]).
* Pregnancy or current breastfeeding.
* Previous eye surgery of any kind.
* Inability to provide informed consent. The ability of the patients in understanding all the aspects of the protocol will be judged by the means of a questionnaire.
* Permanent tattooed makeup (eyeliner, lip, etc.) or general tattoos. Subjects with tattoos will be excluded if those are in a dangerous location in the body or made with colors whose content in iron (e.g. dark blue or dark green) cannot be definitely ruled out by the Investigators.
* Any non-organic implant or any other device such as: cardiac pacemaker, insulin infusion pump, implanted drug infusion device, cochlear, otologic, or ear implant, transdermal medication patch (nitro, hormones) that may cause problems if removed, even temporarily, any metallic implants or objects, body piercing(s), bone/joint pin, screw, nail, plate, wire sutures or surgical staples, shunt.
* Cerebral or other aneurysm clips.
* Shrapnel or other metal imbedded in the patient's body (such as from war wounds or accidents).
* Previous work in metal fields or with machines that may have left any metallic fragments in or near patients' eyes.
* A severe auto accident in the past if it is uncertain that any metal may still be imbedded in the patient's body.
* Any psychological contraindications for MRI (e.g., suffer from claustrophobia). This will be assessed at the time when the medical history will be collected.
* Any contraindications to having study procedures done.

HEALTHY VOLUNTEER INCLUSION CRITERIA:

* Age between 18 and 60.
* Vital signs are found within the normal range at the time of the screening visit.

HEALTHY VOLUNTEER EXCLUSION CRITERIA:

* Clinically significant medical condition that, in the opinion of the investigator, would compromise the patient's safety or affect his/her MRI (e.g., diabetes mellitus, chronic hypertension, severe anemia, kidney disease, heart disease [angina, arrhythmias, congestive heart failure]).
* Pregnancy.
* Previous eye surgery of any kind.
* Inability to provide informed consent.
* Permanent tattooed makeup (eyeliner, lip, etc) or general tattoos. Subjects with tattoos will be excluded if those are in a dangerous location in the body or made with colors (e.g. dark blue and dark green) whose content in iron cannot be definitely ruled out by the Investigators.
* Any non-organic implant or any other device such as: cardiac pacemaker, insulin infusion pump, implanted drug infusion device, cochlear, otologic, or ear implant, transdermal medication patch (Nitro, hormones) that may cause problems if removed even temporarily, any metallic implants or objects, body piercing(s), bone/joint pin, screw, nail, plate, wire sutures or surgical staples, shunt.
* Cerebral or other aneurysm clips.
* Shrapnel or other metal imbedded in the subject's body (such as from war wounds or accidents).
* Previous work in metal fields or with machines that may have left any metallic fragments in or near the subject's eyes.
* A severe auto accident in the past so if it is uncertain whether any metal may still be imbedded in the subject's body.
* Any psychological contraindications for MRI (e.g., suffer from claustrophobia). This will be assessed at the time when the medical history will be collected.
* Any contraindications to having study procedures done.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2006-10-26; Study Completion 2011-09-29

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Noseworthy JH, Lucchinetti C, Rodriguez M, Weinshenker BG. Multiple sclerosis. N Engl J Med. 2000 Sep 28;343(13):938-52. doi: 10.1056/NEJM200009283431307. No abstract available. PMID 11006371
- [Background] Pugliatti M, Rosati G, Carton H, Riise T, Drulovic J, Vecsei L, Milanov I. The epidemiology of multiple sclerosis in Europe. Eur J Neurol. 2006 Jul;13(7):700-22. doi: 10.1111/j.1468-1331.2006.01342.x. PMID 16834700
- [Background] Sospedra M, Martin R. Immunology of multiple sclerosis. Annu Rev Immunol. 2005;23:683-747. doi: 10.1146/annurev.immunol.23.021704.115707. PMID 15771584